CLINICAL TRIAL: NCT05072392
Title: Determining the Effects of Foley Catheter-assisted Nasal Intubation on Nasal Bleeding in Adult Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Eric You-Ten, Associate Professor Anesthesia, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-0005-A
Record Dates: First submitted 2021-10-03; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Nasal Bleeding
Keywords: Endotracheal intubation; Nasal intubation; Epistaxis; Foley catheter; Airway
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Intervention Model Description: Two parallel study groups allocated by randomization to either the intervention group (Foley-assisted nasal endotracheal intubation) or control (standard nasal endotracheal intubation).
  Randomisation is via sealed opaque numbered envelopes that are only opened to reveal group allocation once the patient has been recruited.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to group allocation as they are anesthetised during the intervention procedure.
  The outcome assessor for the primary outcome (incidence of nasal bleeding) will also be blinded by inspecting the gauze swab for blood outside the patient's operating theatre.
  The care provider and investigator are unable to be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley-assisted (Experimental): The tip of the nasal endotracheal tube will be telescoped onto a 16g Foley catheter. If a ballooned catheter is used then the inflation port may be cut off prior to use. The catheter tip is then fed through the pre-selected primary nare, until the tip of the endotracheal tube is in the oropharynx. The catheter is then removed from the tip of the nasal endotracheal tube through the mouth and disposed of. If the nasal endotracheal tube is inappropriately sized, a half size above or below may be used. If difficult to pass, the anesthetist may opt to use the other side nare.
  Following this, the anesthetist will complete the rest of the intubation as usual.
  Interventions: Device: Foley catheter
- Control (No Intervention): The endotracheal tube is passed through the pre-selected primary nare, until the tip of the endotracheal tube is in the oropharynx. If the nasal endotracheal tube is inappropriately sized, a half size above or below may be used. If difficult to pass, the anesthetist may choose to use the other side nare.
  Following this, the anesthetist will complete the rest of the intubation as usual.

INTERVENTIONS:
Device: Foley catheter — Using a 16G Foley catheter to cover the tip of the endotracheal tube as it passes through the nose. This is done in comparison to the standard practice of directly passing an endotracheal tube through the nose without a cover.
  Both groups use warmed endotracheal tubes and the use of topical vasoconstrictor (4 sprays of 0.1% xylometazoline to each nare).
  Arms: Foley-assisted

SUMMARY:
Nasal endotracheal intubation is a well-utilized and important endotracheal intubation route to allow good surgical access for operations involving the oral cavity. Despite its utility, there are potential complications from nasal endotracheal intubation including that of nasal bleeding, which in severe cases can impair the ability to complete the procedure.

The most accepted conventional practice to decrease bleeding associated with nasal endotracheal intubation is to warm the nasal endotracheal tube prior to insertion. However, this technique still yields high rates of nasal bleeding. In 1979, correspondence by MacKinnon and Harrison in Anaesthesia described the use of a flexible urinary catheter (Foley catheter) telescoped onto the endotracheal tube tip to aid atraumatic insertion of the tube. This also served to ensure the tube was not contaminated internally by nasal secretions or blood. This has been more rigorously studied in two RCTs looking at this technique in children, but there has been no similar study in adults.

This study aims to extend the evidence base of the use of this technique in adults. Our hypothesis is that the use of a flexible urinary catheter to telescopically aid nasal intubation will result in a significant decrease in the incidence and severity of nasal bleeding.

DETAILED DESCRIPTION:
The nasal endotracheal intubation technique is an important technique in the management of patients undergoing oral cavity surgery. While usually safe, there are known complications with this technique including nasopharyngeal trauma, epistaxis, bacteremia, endotracheal tube obstruction, retro-pharyngeal perforation, mucosal laceration, olfactory nerve injury, turbinate avulsion, and perforation of the pyriform fossa. There is also a case report of an accidental turbinectomy causing complete obstruction of the endotracheal tube from nasal endotracheal intubation.

As first described in 1979, via correspondence by MacKinnon and Harrison in Anaesthesia, the use of a flexible urinary catheter telescoped onto the endotracheal tube tip can aid atraumatic insertion of a nasal tube and ensure the tube is not contaminated internally by nasal secretions or blood.

This was studied in 2 RCTs in the pediatric population, and both showed a reduction in both the incidence and the severity of bleeding. To the best of our knowledge, there are no RCTs studying the use of a flexible urinary catheter to telescopically aid nasal intubation in the adult population. Thus, the aim of our study is to extend the evidence base for the use of this technique in the adult population. Our hypothesis is that the use of a flexible urinary catheter to telescopically aid nasal intubation will result in statistically and clinically significant reduction in nasal trauma as manifested by bleeding.

Reducing the side effect profile of nasal endotracheal intubation is important to reduce the adverse outcomes from this procedure. Given that the current conventional nasal intubation technique of prewarming the endotracheal tube has high incidence of morbidity i.e. of > 40% incidence of bleeding in adults, and that the flexible urinary catheter to telescopically aid nasal intubation has been shown to decrease the incidence of any bleeding in children when compared to prewarming of the tube, our study will provide further evidence to support regular and ongoing routine use of this technique in adults, which will decrease the morbidity of any patient undergoing this procedure in the future.

40 patients will be randomized to the intervention group (Foley-assisted nasal endotracheal intubation) and 40 patients will be randomized to the control group (standard nasal endotracheal intubation). After obtaining informed written consent and ensuring patients meet the inclusion criteria they will be allocated by the opening of one of the sealed randomization envelopes.

The care-provider anesthetist will have had an email sent out to them beforehand explaining the study protocol, recruitment procedure, flow of the study, and the details of how to perform the Foley catheter assisted nasal intubation technique for the interventional group. Additionally, each care-provider anesthetist assigned to a case for which the patient has provided consent will be contacted the day before the case by a study investigator to remind them of the protocol.

Preoperative care of the patient will be conducted in the usual fashion by the care-provider anesthetist. The care-provider anesthetist will nominate their preferred size of nasal endotracheal tube for their first attempt. 3 nasal endotracheal tube sizes will be prewarmed - the nominated size, plus half a size above and below. Warming will be standardized via placement of the nasal endotracheal tubes in a 1L rigid container of warm saline, left for 15-30 mins in a warming closet set to 43 degrees Celsius. The anesthetist will also nominate the primary nare via which to first attempt intubation. 4 sprays of 0.1% xylometazoline will be administered to each nare prior to induction of general anesthesia.

After induction of general anesthesia, the anesthetist will pass the nasal endotracheal tube of predetermined size through the predetermined nare, until the endotracheal tube tip is present in the oropharynx. The technique for performing this will be based on the group allocation and will either be passed directly through the nose in a standard manner (control group) or will be guided through the nose with a Foley catheter covering the tip (intervention group).

For both groups, if difficulty is encountered entering the oropharynx through the nose then the smaller sized endotracheal tube can be used. For each side, up to three attempts are permitted at passing the endotracheal tube through the nose into the oropharynx. If difficulty is still encountered then the anesthetist may change sides.

Following entry of the endotracheal tube tip into the oropharynx, for both groups, the anesthetist will complete the rest of the intubation as usual. Up to a maximum of 3 attempts at intubation will be permitted. This involves visualization of the glottic opening with a laryngoscope, passage of the tip of the nasal endotracheal tube into the trachea, inflation of the cuff inferior to the vocal cords, confirmation of placement via capnography and clinical signs, and securing the nasal endotracheal tube. A maximum time of 10 minutes is allowed to complete the nasal endotracheal intubation after which the intubation will be recorded as unsuccessful.

If at any point the care-providing anesthetist decides to deviate from the study protocol for patient safety concerns then the trial will be ceased and care will continue as per the care-providing anesthetist. The care-providing anesthetist may also withdraw from the study at any point before or during the procedure in which case the trial will also be ceased.

Data collection and timing will be performed by a study investigator present in the operating theatre.

To measure post-intubation bleeding, the study investigator will perform a swab of the posterior oropharynx. This will be assessed by a different study investigator who will be outside the operating theatre and who will be blinded to group allocation. Degree of bleeding will be graded as no bleeding, trace, moderate, or severe according to the scale from EA Algadiem et al.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Scheduled to undergo an operation requiring nasotracheal intubation

Exclusion Criteria:

* Latex allergy
* Emergency surgery
* High risk of aspiration
* Anticipated or unanticipated difficult airway or bag mask ventilation
* Morbid obesity (BMI >40)
* Bleeding diathesis
* Basal skull fracture
* Previous deviated nasal septum surgery
* Nasal polyps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-04 (Estimated); Primary Completion 2022-05-14 (Estimated); Study Completion 2022-05-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of nasal bleeding | 10 minutes (must be assessed prior to surgical start as this may cause additional bleeding)
  Defined as the presence of blood on a folded stack of two 4x4 inch gauze swabs to the posterior oropharynx after the confirmation of successful nasotracheal intubation

SECONDARY OUTCOMES:
Severity of bleeding | 10 minutes (must be assessed prior to surgical start as this may cause additional bleeding)
  Defined as trace, moderate, or severe bleeding by comparing gauze saturation to referenced illustrations from EA Algadiem et al. whereby trace bleeding is defined as blood present but <25% gauze saturation (or 3mL of blood), moderate bleeding is 25% gauze saturation (or 3mL of blood) and severe bleeding is 50% gauze saturation (or 6mL of blood)
Time to successful intubation | 10 minutes
  Defined as time in seconds from when the endotracheal tube is first inserted into the nare until the presence of an end-tidal capnography waveform
Number of attempts at intubation | 10 minutes
  Defined as the number of times a laryngoscope is inserted into the patient's mouth
Incidence of requirement to suction blood from the oral cavity to facilitate intubation | 10 minutes
  Defined as the requirement of the care-provider anesthetist to use a yankauer suction device to suction blood from the airway prior to obtaining an end-tidal capnography waveform
Incidence of significant postop nasal bleeding | 24 hours
  Defined as the presence of nasal bleeding requiring intervention (such as compression packing or vasoconstrictor agents) between the end of the surgical procedure and when the patient leaves the post-anaesthesia care unit (PACU/recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Kong Eric You-Ten, MD PhD FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underlie results in a publication. All data will be deidentified and will be referenced using their study participant number.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication

REFERENCES:
- [Background] Ali Algadiem E, Aleisa AA, Alsubaie HI, Buhlaiqah NR, Algadeeb JB, Alsneini HA. Blood Loss Estimation Using Gauze Visual Analogue. Trauma Mon. 2016 May 3;21(2):e34131. doi: 10.5812/traumamon.34131. eCollection 2016 May. PMID 27626017